CLINICAL TRIAL: NCT02060201
Title: A Bioequivalence Study of 2.5-mg Saxagliptin/5-mg Dapagliflozin and 5-mg Saxagliptin/10-mg Dapagliflozin Fixed Dose Combination Tablets Relative to Coadministration of Their Respective Individual Components in Healthy Subjects and a Characterization of the Effect of Food on the Fixed Dose Combination Tablets
Brief Title: Bioequivalence/Food Effect - Saxa/Dapa Dual Fixed Dose Combination (FDC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-341; 118,840 (Other: IND Number)
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A: Saxagliptin 2.5mg+Dapagliflozin 5mg; Fasting (Other): Saxagliptin 2.5 mg tablet and Dapagliflozin 5 mg tablet single dose orally on Day 1 in one of 3 periods
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- Treatment B: Saxagliptin 2.5mg/Dapagliflozin 5mg FDC; Fasting (Other): Saxagliptin 2.5 mg/Dapagliflozin 5 mg fixed dose combination tablet single dose orally on Day 1 in one of 3 periods
  Interventions: Drug: Saxagliptin/Dapagliflozin FDC
- Treatment C: Saxagliptin 2.5mg/Dapagliflozin 5mg FDC; Fed (Other): Saxagliptin 2.5 mg/Dapagliflozin 5 mg fixed dose combination tablet single dose orally on Day 1 in one of 3 periods
  Interventions: Drug: Saxagliptin/Dapagliflozin FDC
- Treatment D: Saxagliptin 5mg+Dapagliflozin 10mg; Fasting (Other): Saxagliptin 5 mg tablet and Dapagliflozin 10 mg tablet single dose orally for on Day 1 in one of 3 periods
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- Treatment E: Saxagliptin 5mg/Dapagliflozin 10mg FDC; Fasting (Other): Saxagliptin 5 mg/Dapagliflozin 10 mg fixed dose combination tablet single dose orally on Day 1 in one of 3 periods
  Interventions: Drug: Saxagliptin/Dapagliflozin FDC
- Treatment F: Saxagliptin 5mg/Dapagliflozin 10mg FDC; Fed (Other): Saxagliptin 5 mg/Dapagliflozin 10 mg fixed dose combination tablet single dose orally on Day 1 in one of 3 periods
  Interventions: Drug: Saxagliptin/Dapagliflozin FDC

INTERVENTIONS:
Drug: Saxagliptin
  Other Names: Onglyza®; BMS-477118
  Arms: Treatment A: Saxagliptin 2.5mg+Dapagliflozin 5mg; Fasting; Treatment D: Saxagliptin 5mg+Dapagliflozin 10mg; Fasting
Drug: Dapagliflozin
  Other Names: Farxiga®; Forxiga®; BMS-512148
  Arms: Treatment A: Saxagliptin 2.5mg+Dapagliflozin 5mg; Fasting; Treatment D: Saxagliptin 5mg+Dapagliflozin 10mg; Fasting
Drug: Saxagliptin/Dapagliflozin FDC
  Other Names: BMS-986098
  Arms: Treatment B: Saxagliptin 2.5mg/Dapagliflozin 5mg FDC; Fasting; Treatment C: Saxagliptin 2.5mg/Dapagliflozin 5mg FDC; Fed; Treatment E: Saxagliptin 5mg/Dapagliflozin 10mg FDC; Fasting; Treatment F: Saxagliptin 5mg/Dapagliflozin 10mg FDC; Fed

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence (BE) of Saxagliptin and Dapagliflozin from a 2.5-mg Saxagliptin/5-mg Dapagliflozin FDC tablet after oral administration relative to 2.5-mg Saxagliptin and 5-mg Dapagliflozin tablets administered orally together in the fasted state and to demonstrate the BE of Saxagliptin and Dapagliflozin from a 5-mg Saxagliptin/10-mg Dapagliflozin FDC tablet after oral administration relative to 5-mg Saxagliptin and 10-mg Dapagliflozin tablets administered orally together in the fasted state. Demonstrating bioequivalence refers to showing that the FDC tablet and co-administration of the individual components yield similar blood levels/concentrations of the drug and are handled by the body similarly.

DETAILED DESCRIPTION:
Primary Purpose: This study is designed to demonstrate the bioequivalence of Saxagliptin and Dapagliflozin from a FDC tablet after oral administration relative to Saxagliptin and Dapagliflozin tablets administered orally together in the fasted and fed state

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination (PE), vital signs, 12-lead ECG, and clinical laboratory determinations
* Body mass index (BMI) of 18.5 to 30 kg/m(2)
* Men and women, ages 18 to 50 years
* Women of childbearing potential must use acceptable methods of highly effective birth control

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* History of chronic or recurrent urinary tract infection for females
* History of glucose intolerance or diabetes mellitus
* History of allergies or adverse reactions to Dipeptidyl peptidase-IV (DPP4) or Sodium-glucose cotransporter (SGLT) inhibitors
* Prior exposure to Saxagliptin or Dapagliflozin or related drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin and 42 time points for Dapagliflozin up to 15 days
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [(AUC(0-T)] for Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin and 42 time points for Dapagliflozin up to 15 days
Area under the concentration-time curve from time zero extrapolated to infinite time [(AUC(INF)] for Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin and 42 time points for Dapagliflozin up to 15 days

SECONDARY OUTCOMES:
Cmax for 5-hydroxy (OH) Saxagliptin | 54 time points up to 15 days
AUC(0-T) for 5-hydroxy (OH) Saxagliptin | 54 time points up to 15 days
AUC(INF) for 5-hydroxy (OH) Saxagliptin | 54 time points up to 15 days
Time of maximum observed plasma concentration (Tmax) for Saxagliptin, 5-OH Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin, 5-OH Saxagliptin and 42 time points for Dapagliflozin up to 15 days
Percent of AUC extrapolated from last quantifiable concentration to infinity (pAUCe) for Saxagliptin, 5-OH Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin, 5-OH Saxagliptin and 42 time points for Dapagliflozin up to 15 days
Half life (T HALF) for Saxagliptin, 5-OH Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin, 5-OH Saxagliptin and 42 time points for Dapagliflozin up to 15 days
Terminal disposition rate constant (Lambda) for Saxagliptin, 5-OH Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin, 5-OH Saxagliptin and 42 time points for Dapagliflozin up to 15 days
Time point where log-linear elimination begins (TLIN) for Saxagliptin, 5-OH Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin, 5-OH Saxagliptin and 42 time points for Dapagliflozin up to 15 days
Time at which the last concentration occurred that is above the lower limit of quantitation (LQCT) for Saxagliptin, 5-OH Saxagliptin and Dapagliflozin | 54 time points for Saxagliptin, 5-OH Saxagliptin and 42 time points for Dapagliflozin up to 15 days
Safety measured by the occurrence of deaths, adverse events (AEs), serious adverse events (SAEs), results of clinical laboratory tests, vital sign measurements, physical examination findings, and 12-lead electrocardiogram (ECG) results | Approximately up to 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb